CLINICAL TRIAL: NCT06360419
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Solriamfetol in Subjects With Major Depressive Disorder
Brief Title: Progressing TAAR-1, Dopamine, and Norepinephrine in Depression Using Solriamfetol
Acronym: PARADIGM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOL-MDD-301
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: Solriamfetol; Sunosi; MDD; Major Depressive Disorder; Axsome; Non-stimulant therapy; Dopamine norepinephrine reuptake inhibitor; Trace amine-associated receptor 1 (TAAR1) agonist
MeSH Terms: conditions — Depressive Disorder, Major | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solriamfetol 300 mg (Experimental): Up to 6 weeks
  Interventions: Drug: Solriamfetol 300 mg
- Placebo (Placebo Comparator): Up to 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol 300 mg — Solriamfetol tablets, taken once daily
  Arms: Solriamfetol 300 mg
Drug: Placebo — Placebo tablets, taken once daily
  Arms: Placebo

SUMMARY:
PARADIGM (Progressing TAAR-1, Dopamine, and Norepinephrine in Depression Using Solriamfetol) is a Phase 3, randomized, double-blind, placebo-controlled, multicenter trial to assess the safety and efficacy of solriamfetol for the treatment of major depressive disorder (MDD) in adults.

DETAILED DESCRIPTION:
Eligible subjects must have a primary diagnosis of MDD without psychotic features based on the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria. Subjects will be randomized in a 1:1 ratio to receive either solriamfetol (300 mg) or placebo for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Currently meets the DSM-5 criteria for MDD without psychotic features, based on the SCID-5-CT
* Current major depressive episode
* Male or female, aged 18 to 65 inclusive

Exclusion Criteria:

* Prior exposure to solriamfetol/Sunosi, through either a clinical study or prescription
* Unable to comply with study procedures
* Medically inappropriate for study participation in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 weeks
Incidence of treatment-emergent adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Bellflower, California
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Lemon Grove, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Montclair, California
  - Clinical Research Site, Oceanside, California
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Riverside, California
  - Clinical Research Site, Sherman Oaks, California
  - Clinical Research Site, Torrance, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, Cromwell, Connecticut
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site, Overland Park, Kansas
  - Clinical Research Site, New Orleans, Louisiana
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Saint Charles, Missouri
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Media, Pennsylvania
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Friendswood, Texas
  - Clinical Research Site, Wichita Falls, Texas
  - Clinical Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com